CLINICAL TRIAL: NCT06521710
Title: Phase I Clinical Trial: Pilot Study of Intraoperative Somatic-Autonomic Nerve Grafting Technique to Preserve Erectile Function in Patients With High Grade Prostate Cancer Undergoing Robotic Assisted Radical Prostatectomy
Brief Title: Nerve Grafting Technique to Preserve Erectile Function in Patients Undergoing Robotic Assisted Radical Prostatectomy
Acronym: NR-RALP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Victor McPherson, MD, MSc, FRCSC, Assistant Professor Division of Urology, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-4129
Record Dates: First submitted 2024-07-21; First posted 2024-07-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer; Erectile Dysfunction
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NR-RALP (Experimental): Nerve Grafting Technique in patients with High Grade Prostate Cancer Undergoing Robotic Assisted Radical Prostatectomy
  Interventions: Procedure: Intraoperative Somatic-Autonomic Nerve Grafting

INTERVENTIONS:
Procedure: Intraoperative Somatic-Autonomic Nerve Grafting — A one-sided graft using a genitofemoral (GFN) nerve graft between one obturator nerve and the corpora cavernosa

SUMMARY:
The investigator proposing a single arm prospective pilot trial evaluating the safety and the 1-year erectile recovery outcomes of patients undergoing Nerve Restoring (NR) Robotically assisted laparoscopic radical prostatectomy (RALP). During this study a total of 10 patients who are undergoing robotic prostatectomy will have their surgery performed utilizing a novel technique, NR-RALP, which incorporates a genitofemoral (GFN) nerve graft designed to try to improve the erectile function and recovery of men undergoing standard of care robotic prostatectomy while minimizing additional morbidity of the procedure

DETAILED DESCRIPTION:
Patients will have baseline evaluation with International Index of Erectile Function-5 (IIEF-5) questionnaire and the Short Form McGill Pain Questionnaire (SF-MPQ)1, which will be re-evaluation at time of their standard of care post-operative visits at 4 weeks, 3-, 6-, 12- and 18-months. Post-operative safety will be assessed by recording any clinically detected complications during their peri- and post-operative care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing standard of care robotic radical prostatectomy for high-risk localized prostate cancer as defined by any of:

   1. Gleason grade ≥8
   2. PSA ≥20
   3. >pT2 on preoperative MRI imaging
2. Patients must have preoperative erectile function with a baseline IIEF score of ≥17

Exclusion Criteria:

1. Patients with previous pelvic surgery
2. Patients with previous pelvic radiotherapy
3. Patient with previous focal therapy for prostate cancer
4. Patients aged < 18 years at diagnosis
5. Legally incapable patients
6. Patients who are unable to complete questionnaires and have no companion to help complete them
7. Patients undergoing a concomitant cancer surgery
8. Patients with pre-existing neurologic disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events measured by the Clavian-Dindo classification | Through study completion, an average of 18 months
  The primary outcome is specifically the safety of the operation measured by adverse events as defined by the Clavian-Dindo classification. The measurement varies from Grade I (Best possible outcome) to Grade V (Worst possible outcome).
  Grade I Deviation from normal p/o course. No pharmacological or surgical treatment, endoscopic or radiological interventions were required. Acceptable therapeutic drugs such as anti-emetics, antipyretics, analgesics, diuretics,electrolytes, physiotherapy. Wound infections, small abscess requiring incision at bedside.
  Grade II Normal course altered. Pharmacological management other than in Grade I. Blood transfusions and total parenteral nutrition are also included.
  Grade III Complications that require intervention of various degrees. Grade IV Complications threatening life of patients (including Central Nervous System complications), requiring Intensive Treatment Unit support.
  Grade V Death of a patient.

SECONDARY OUTCOMES:
International Index of Erectile Function-5 (IIEF-5) | Screening pre-NR-RALP procedure
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool.
  Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 4-6 weeks post-NR-RALP procedure
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool.
  Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 3 months post-NR-RALP procedure
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool.
  Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 6 months post-NR-RALP procedure
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool.
  Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 12 months post-NR-RALP procedure
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool.
  Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 18 months post-NR-RALP procedure
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool.
  Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
Short Form McGill Pain Questionnaire (SF-MPQ) | Screening pre-NR-RALP procedure
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
  The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 4-6 weeks post-NR-RALP procedure
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
  The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 3 months post-NR-RALP procedure
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
  The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 6 months post-NR-RALP procedure
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
  The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 12 months post-NR-RALP procedure
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
  The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 18 months post-NR-RALP procedure
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
  The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Victor McPherson, MD, Principal Investigator — Jewish General Hospital
Locations (2):
- Canada (2):
  - Jewish General Hospital, CIUSSS Centre-Ouest de l'île de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec